CLINICAL TRIAL: NCT03891979
Title: A Pilot Study of Gut Microbiome Modulation to Enable Efficacy of Checkpoint-based Immunotherapy in Pancreatic Adenocarcinoma
Brief Title: Gut Microbiome Modulation to Enable Efficacy of Checkpoint-based Immunotherapy in Pancreatic Adenocarcinoma
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Suspended due to Primary Investigator's decision
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-00137
Record Dates: First submitted 2019-03-25; First posted 2019-03-27 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — pembrolizumab; Ciprofloxacin; Metronidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab + Antibiotics (Experimental): Pembrolizumab will be given for two doses every 3 weeks starting on day 8 (ie days 8 and 29). Antibiotics will continue throughout the entire four week pre-operative period.
  Interventions: Drug: Pembrolizumab; Drug: Ciprofloxacin 500mg PO BID days 1-29; Drug: Metronidazole 500mg PO TID days 1-29

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab will be given for two doses every 3 weeks starting on day 8 (ie days 8 and 29). Antibiotics will continue throughout the entire four week pre-operative period.
  Ciprofloxacin 500mg PO BID days 1-29; Metronidazole 500mg PO TID days 1-29; Pembrolizumab 200mg IV days 8 and 29.
Drug: Ciprofloxacin 500mg PO BID days 1-29 — Antibiotics will continue throughout the entire four week pre-operative period.
Drug: Metronidazole 500mg PO TID days 1-29 — Antibiotics will continue throughout the entire four week pre-operative period.

SUMMARY:
A multi-institutional, single arm pilot study of antibiotics and pembrolizumab for the treatment of surgically resectable pancreatic cancer. The primary purpose of this study is to determine the change in immune activation in pancreatic tumor tissue following treatment with antibiotics and pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed pancreatic adenocarcinoma. Histologies other than adenocarcinoma, or any mixed histologies, will NOT be eligible. *Note: histology must be confirmed prior to study treatment, however, participants may be consented to study based on imaging results consistent with pancreatic adenocarcinoma and then undergo diagnostic and research biopsy simultaneously.
* Clinical stage I and II disease (per AJCC 8th ed)
* Resectable pancreatic cancer as defined by NCCN Guidelines 1.2018 and based on pancreatic protocol dual-phase CT imaging. Multi-detector computed tomography (MDCT) angiography, performed by acquiring thin, preferably sub-millimeter, axial sections using a dual-phase pancreatic protocol, with images obtained in the pancreatic and portal venous phase of contrast enhancement, is required.
* No arterial tumor contact (celiac axis [CA], superior mesenteric artery [SMA], or common hepatic artery [CHA])
* No tumor contact with the superior mesenteric vein (SMV) or portal vein (PV) or ≤180° contact without vein contour irregularity
* Patients must agree to pre-treatment biopsy and definitive surgical resection
* ECOG performance status of 0 or 1
* No prior treatment for diagnosis of pancreatic cancer
* Normal organ and marrow function
* Absolute neutrophil count (ANC) ≥1500/µL
* Platelets ≥100 000/µL
* Hemoglobin ≥9.0 g/dL or ≥5.6 mmol/La
* Renal Creatinine OR Measured or calculated by creatinine clearance (GFR can also be used in place of creatinine or CrCl) ≤1.5 × ULN OR

  ≥30 mL/min for participant with creatinine levels >1.5 × institutional ULN
* Hepatic Total bilirubin ≤1.5 ×ULN OR direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN
* AST (SGOT) and ALT (SGPT) ≤2.5 × ULN
* Coagulation International normalized ratio (INR) OR prothrombin time (PT)
* Activated partial thromboplastin time (aPTT) ≤1.5 × ULN unless participant is receiving anticoagulant therapy as long as PT or aPTT is within therapeutic range of intended use of anticoagulants
* ALT (SGPT)=alanine aminotransferase (serum glutamic pyruvic transaminase); AST (SGOT)=aspartate aminotransferase (serum glutamic oxaloacetic transaminase); GFR=glomerular filtration rate; ULN=upper limit of normal.
* Criteria must be met without erythropoietin dependency and without packed red blood cell (pRBC) transfusion within last 2 weeks.
* Creatinine clearance (CrCl) should be calculated per institutional standard. Note: This table includes eligibility-defining laboratory value requirements for treatment; laboratory value requirements should be adapted according to local regulations and guidelines for the administration of specific chemotherapies.
* Ability to understand and sign a written informed consent document. Participant must have willingness and ability to comply with scheduled visits, treatment plans, laboratory tests and other study procedures.
* A female participant is eligible to participate if she is not pregnant (see Appendix 1), not breastfeeding, and at least one of the following conditions applies:
* Not a woman of childbearing potential (WOCBP) as defined in Appendix 1 OR
* A WOCBP who agrees to follow the contraceptive guidance in Appendix 1 during the treatment period and for at least 120 days plus 30 days (a menstruation cycle) after the last dose of study treatment.
* Males who are sexually active with WOCBP must agree to follow instructions for method(s) of contraception (see Appendix 1) for the duration of treatment with study treatment(s) and for a total of 180 days posttreatment completion. In addition, male participants must be willing to refrain from sperm donation during this time.

Exclusion Criteria:

* Borderline resectable, locally advanced or distant metastatic disease
* Any medical condition which makes definitive surgical resection of the pancreatic cancer contraindicated due to high risk of morbidity/mortality
* Has active autoimmune disease that has required systemic treatment in past 2 years (ie, with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment.

  4. Medical history and concurrent disease as below:

  • Participants with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalents) or other immunosuppressive medications within 14 days of study treatment administration except for adrenal replacement steroid doses > 10 mg daily prednisone equivalent in the absence of active autoimmune disease.

Note: Treatment with a short course of steroids (< 5 days) up to 7 days prior to initiating study treatment is permitted. Participants with asthma that require intermittent use intermittent use of bronchodilators, inhaled steroids, or local steroid injections would not be excluded from the study.

* Interstitial lung disease that is symptomatic or may interfere with the detection or management of suspected treatment-related pulmonary toxicity.
* Uncontrolled or significant cardiovascular disease including, but not limited to, any of the following:

  * Myocardial infarction or stroke/transient ischemic attack within the past 6 months
  * Uncontrolled angina within the past 3 months
  * Any history of clinically significant arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes)
  * History of other clinically significant heart disease (eg, cardiomyopathy, congestive heart failure with New York Heart Association functional classification III to IV, pericarditis, significant pericardial effusion, or myocarditis)
  * Cardiovascular disease-related requirement for daily supplemental oxygen therapy.
* Evidence of uncontrolled, active infection, requiring parenteral or oral anti-bacterial, anti-viral or anti-fungal therapy ≤ 28 days prior to screening on study.
* Participants with a condition requiring chronic systemic oral treatment with either antibiotics or anti-fungals
* Any uncontrolled inflammatory GI disease including Crohn's Disease and ulcerative colitis.

  * Participants with active, known, or suspected autoimmune disease. Participants with vitiligo, type I diabetes mellitus, residual hypothyroidism due to autoimmune condition only requiring hormone replacement, euthyroid participants with a history of Grave's disease (participants with suspected autoimmune thyroid disorders must be negative for thyroglobulin and thyroid peroxidase antibodies and thyroid stimulating immunoglobulin prior to first dose of study treatment), psoriasis not requiring systemic treatment, or conditions not expected to recur in the absence of an external trigger are permitted to enroll after discussing with the Principal Investigator.
  * Has received a live vaccine within 30 days prior to the first dose of study drug. Examples of live vaccines include, but are not limited to, the following: measles, mumps, rubella, varicella/zoster (chicken pox), yellow fever, rabies, Bacillus Calmette-Guérin (BCG), and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (eg, FluMist®) are live attenuated vaccines and are not allowed. *Note: for those participants who will be undergoing planned splenectomy, vaccinations against S. pneumoniae, N. meningitidis, H. influenzae type b and influenza virus should be administered at least 2 weeks after the surgical intervention.
  * Known human immunodeficiency virus (HIV), known active hepatitis A, or known hepatitis B or C infection.
  * History of acute diverticulitis within the last 6 months or current chronic diarrhea
  * Expected to require any other form of antineoplastic or surgical therapy while on study
  * Pregnant or lactating women
  * A WOCBP who has a positive urine pregnancy test within 72 hours or no pregnancy test prior to registration (see Appendix 1). If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.

Note: in the event that >72 hours have elapsed between the screening pregnancy test and the first dose of study treatment, another pregnancy test (urine or serum) must be performed and must be negative in order for subject to start receiving study medication.

* WOCBP who are unwilling or unable to use an acceptable method to minimize the risk of pregnancy (see Appendix 1) for the entire study period and 120 days plus 30 days (a menstruation cycle) after the last dose of study treatment. WOCBP who are continuously not heterosexually active are also exempt from contraceptive requirements, but still must undergo pregnancy testing as described in section 20.
* Sexually active fertile men not using effective birth control if their partners are WOCBP
* History of primary immunodeficiency
* Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
* History of organ allograft or allogeneic bone marrow transplant.
* Any prior radiation therapy, immunotherapy, or biologic ('targeted') therapy for treatment of the patient's pancreatic tumor. Biliary stent is allowed.
* Treatment for other invasive carcinomas within the last two years who are at greater than 5% risk of recurrence at time of eligibility screening. Carcinoma in-situ and basal cell carcinoma/ squamous cell carcinoma of the skin are allowed.
* Participation in any investigational drug study within 4 weeks preceding the start of study treatment.
* Major surgery, excluding laparoscopy, within 4 weeks of the start of study treatment, without complete recovery.
* History of allergy to study treatments or any of its components

Ages: 18 Months to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-06-25 (Actual); Primary Completion 2020-06-01 (Actual); Study Completion 2020-06-01 (Actual)

PRIMARY OUTCOMES:
Change in immune activation in pancreatic tumor tissue following treatment with antibiotics and pembrolizumab measured by activation of HLA-DR, | 12 Weeks
  activation is defined as an increase of 20% or more over baseline in percentage of T cells expressing the marker.
Change in immune activation in pancreatic tumor tissue following treatment with antibiotics and pembrolizumab measured by activation of | 12 Weeks
  activation is defined as an increase of 20% or more over baseline in percentage of T cells expressing the marker.

CONTACTS AND LOCATIONS:
Overall Officials: Deidre Cohen, Principal Investigator — New York Langone Medical Center
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after deidentification (text, tables, figures, and appendices).
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research.
Access Criteria: Upon reasonable request. Requests should be directed to Kirsten.Swingle@nyulangone.org. To gain access, data requestors will need to sign a data access agreement